CLINICAL TRIAL: NCT06046729
Title: A Phase 2b, Double-Blind, Placebo-Controlled Study to Evaluate Eltrekibart in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study of Eltrekibart (LY3041658) in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18518; I7P-MC-DSAF (Other: Eli Lilly and Company); 2023-505608-43-00 (Other: EU Trial Number); U1111-1292-6255 (Other: UTN Number)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Phase 2b
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Eltrekibart Dose 1 (Experimental): Eltrekibart will be given subcutaneously (SC).
  Interventions: Drug: Eltrekibart
- Eltrekibart Dose 2 (Experimental): Eltrekibart will be given SC.
  Interventions: Drug: Eltrekibart
- Eltrekibart Dose 3 (Experimental): Eltrekibart will be given SC.
  Interventions: Drug: Eltrekibart
- Placebo (Placebo Comparator): Placebo will be given.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrekibart — Administered SC
  Other Names: LY3041658
  Arms: Eltrekibart Dose 1; Eltrekibart Dose 2; Eltrekibart Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This study aims to find the appropriately safe and effective dose and dosing frequency for eltrekibart in adults with moderate-to-severe hidradenitis suppurativa (HS) for further clinical development. The study will last approximately 62 weeks and may include up to 31 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HS for at least 12 months.
* Have HS lesions in at least 2 distinct anatomical regions. At least 1 of the lesions must be at least Hurley Stage II or III.
* Have an (abscess plus inflammatory nodule) count of at least 5.
* Agree to use topical antiseptics daily.
* Had an inadequate response or intolerance to a 28-day course of oral antibiotics.

Exclusion Criteria:

* Have more than 20 draining fistulae.
* Have had surgical treatment for HS in the last 4 weeks before randomization.
* Have an active skin disease or condition, that could interfere with the assessment of HS.
* Have a current or recent acute, active infection.
* Are immunocompromised.
* Have a history of chronic alcohol abuse, IV drug abuse, or other illicit drug abuse within 1 year before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participant Achieving Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) | Week 16

SECONDARY OUTCOMES:
Mean Change from Baseline in Total Number of Abscesses and Inflammatory Nodules | Baseline, Week 16
Mean Change from Baseline in HS-related Average Skin Pain Numerical Rating Scale (NRS) | Baseline, Week 16
Pharmacokinetics (PK): Plasma Concentrations of Eltrekibart | Baseline through Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (74):
- United States (42):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Saguaro Dermatology Associates, LLC - Probity - PPDS, Phoenix, Arizona
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Institute and Skin Care Center, Santa Monica, California
  - University of Connecticut, Farmington, Connecticut
  - Direct Helpers Research Center, Hialeah, Florida
  - University of Miami, Miami, Florida
  - Skin Research of South Florida, Miami, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Advanced Medical Research, PC, Sandy Springs, Georgia
  - NorthShore Medical Group Dermatology - Skokie, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Equity Medical - Bowling Green, Bowling Green, Kentucky
  - Derm Research LLC, Louisville, Kentucky
  - Care Access-Marriottsville, Marriottsville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Revival Research Institute - Troy, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Skin Specialists, P.C, Omaha, Nebraska
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - Darst Dermatology, Charlotte, North Carolina
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - DermDox Centers for Dermatology, Camp Hill, Pennsylvania
  - DermDox Dermatology Centers, Sugarloaf, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Columbia Dermatology & Aesthetics, Columbia, South Carolina
  - International Clinical Research - Tennessee (IC Research), Murfreesboro, Tennessee
  - Advanced Research Experts, Nashville, Tennessee
  - Modern Research Associates, Dallas, Texas
  - North Texas Clinical Research, Frisco, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Dermatology Specialists of Spokane, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - East Sydney Doctors, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Sinclair Dermatology - East Melbourne, East Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Holdsworth House Medical Practice, Sydney
- Canada (7):
  - Beacon Dermatology, Calgary, Alberta
  - Alberta Dermasurgery Centre, Edmonton, Alberta
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Brunswick Dermatology Center, Fredericton, New Brunswick
  - Simcoderm Medical & Surgical Dermatology Centre, Barrie, Ontario
  - DermEffects - Probity - PPDS, London, Ontario
  - Center de Recherche St Louis, Québec, Quebec
- Germany (8):
  - Hautklinik Erlangen, Erlangen, Bavaria
  - Hautarztpraxis Mahlow, Blankenfelde-Mahlow, Brandenburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitaetsklinikum der Ruhr-Universitaet Bochum (UKRUB) - St. Josef-Hospital, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, Westfalen
  - Hautzentrum Friedrichshain - Dermatologie, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Greece (3):
  - Hospital of Venereal and Skin Diseases A.Syggros, Athens, Attica
  - University General Hospital of Heraklion Loc. 1, Heraklion, Irakleío
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki, Thessaloníki
- Poland (7):
  - Cityclinic Przychodnia Lekarsko Psychologiczna Matusiak Spółka Partnerska, Wroclaw, Lower Silesian Voivodeship
  - Wro Medica, Wroclaw, Lower Silesian Voivodeship
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Klinika Badawcza Centrum Badan Klinicznych Wojciech Brzezicki, Malbork, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - Dermoklinika-Centrum Medyczne s.c, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Eltrekibart (LY3041658) in Adult Participants With Moderate to Severe Hidradenitis Suppurativa — https://trials.lilly.com/en-US/trial/424355